CLINICAL TRIAL: NCT04027374
Title: Epigenetic Alterations in Stress Regulation Genes Among Newborns After Fetal Surgery for Myelomeningocele Repair: An Exploratory Study
Brief Title: Stress-associated Epigenetic Alterations in Newborns After Fetal Surgery
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Zurich (Other); Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2019-00598
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Meningomyelocele
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA sample collection from the child will take place between 24 and 72 hours of life during hospitalization by trained research project staff. In order to obtain DNA and RNA, saliva will be collected using special sponge devices designed for use with infants who cannot spit independently.
  For DNA, 2x ORAcollect for pediatrics (OC-175; DNA Genotek Inc) will be used to collect saliva in order to obtain enough DNA sample.
  For RNA, 2x saliva collection devices for pediatrics (CP-190; DNA Genotek Inc) will be used to collect saliva in order to obtain enough RNA sample from the newborns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fetal surgery group: Newborns after successful fetal surgery for MMC, delivered by elective c-section at weeks 35;0 - 37;0.
  Interventions: Procedure: Fetal surgery for MMC repair
- Glucocorticoid control group: Healthy newborns after exposure to synthetic glucocorticoids for lung maturity during pregnancy, delivered by elective c-section between 35;0 - 40;0 weeks, matched for child sex with group 1. This group is needed to control for the effects of sGC exposure.
- Healthy controls: Healthy newborns, uncomplicated pregnancy, delivered at term by elective c-section between 36;0 - 39;0 weeks. Matched for child sex with group 1.

INTERVENTIONS:
Procedure: Fetal surgery for MMC repair — Fetal surgery for MMC repair
  Groups: Fetal surgery group

SUMMARY:
Open spina bifida or myelomeningocele (MMC) is a devastating congenital defect of the central nervous system for which there is no cure. The etiology of MMC remains poorly understood. Primary failure of neural tube closure at the caudal neuropore in the embryonic period results in exposure of the developing spinal cord to the uterine environment. Without protective tissue coverage, secondary destruction of the exposed neural tissue by trauma or amniotic fluid may occur throughout gestation. In order to protect the spinal cord from this secondary destruction, a fetal surgical repair can be performed between gestational weeks 20 and 26.

From a psychological point of view fetal repair of MMC constitutes a highly stressful event both for the mother and the fetus. To date, however, stress of mothers and children in case of prenatal surgery for MMC repair has never been studied. It is therefore unclear, if and to what extend the procedure and its consequences are associated with stress, and if there are short- or longer-term consequences.

The aims of this study are threefold:

1. Do newborns after fetal surgery for MMC show epigenetic alterations in genes that are involved in stress regulation?
2. With which medical and psychosocial variables are epigenetic alterations associated?
3. At age 3 months, do infants after fetal surgery have a more difficult temperament compared to controls?

DETAILED DESCRIPTION:
BACKGROUND AND AIMS:

Open spina bifida or myelomeningocele (MMC) is a devastating congenital defect of the central nervous system for which there is no cure. The etiology of MMC remains poorly understood. Primary failure of neural tube closure at the caudal neuropore in the embryonic period results in exposure of the developing spinal cord to the uterine environment. Without protective tissue coverage, secondary destruction of the exposed neural tissue by trauma or amniotic fluid may occur throughout gestation. In order to protect the spinal cord from this secondary destruction, a fetal surgical repair can be performed between gestational weeks 20 and 26.

From a psychological point of view fetal repair of MMC constitutes a highly stressful event both for the mother and the fetus. To date, however, stress of mothers and children in case of prenatal surgery for MMC repair has never been studied. It is therefore unclear, if and to what extend the procedure and its consequences are associated with stress, and if there are short- or longer-term consequences.

The aims of this study are threefold:

1. Do newborns after fetal surgery for MMC show epigenetic alterations in genes that are involved in stress regulation?
2. With which medical and psychosocial variables are epigenetic alterations associated?
3. At age 3 months, do infants after fetal surgery have a more difficult temperament compared to controls?

METHODS:

Sample: The study will include newborns after fetal surgery for MMC at the University Hospital Zurich and two control groups. One including healthy newborns and another including newborns after prenatal exposure to synthetic glucocorticoids (sGC) in pregnancy. Each group shall include n=30 newborns (i.e. total number of study participants: n=90).

Recruitment and Procedures: Recruitment will take place at the University Children's Hospital and the University Hospital Zürich and will be continued until the required sample size is reached. For every MMC-patient, secondary recruitment of a control child for group 2 and 3 will be performed (matched for child sex). Parents of all study groups will be approached by the responsible study staff after checking for inclusion and exclusion criteria. They will be informed orally about the study and the study information letter (see encl.) will be provided. Parents will be contacted again after >24h face to face or by phone by study staff to answer any questions, if necessary. If the parents agree to participate in the study, they will provide the signed written informed consent form (see encl.). After inclusion in the study, the parents will be contacted again in hospital by study staff around 24-36 hours after birth to re-explain the collection of the saliva samples. The saliva samples will then be collected between 24 and 72h postpartum. Six weeks and 3 months post-partum, the parents will receive the study questionnaires by mail and they will be asked to complete and return them within 1 week. If the questionnaires are not received after 10 days, study staff will contact the parents by phone for a gentle reminder. Parents are not financially compensated for taking part in the study.

Collected data:

-) DNA and RNA sample collection from the child will take place between 24 and 72 hours of life during hospitalization by trained research project staff. In order to obtain DNA and RNA, saliva will be collected using special sponge devices designed for use with infants who cannot spit independently.

For DNA, 2x ORAcollect for pediatrics (OC-175; DNA Genotek Inc) will be used to collect saliva in order to obtain enough DNA sample.

For RNA, 2x saliva collection devices for pediatrics (CP-190; DNA Genotek Inc) will be used to collect saliva in order to obtain enough RNA sample from the newborns.

* Medical data: a) Child: Gestational age at birth; gender; birth length and percentile; birth weight and percentile; head circumference at birth and percentile; Apgar score; umbilical artery ph and lactate; meconium-stained amniotic fluid; Gestational age at fetal surgery; time and length of fetal surgery; positioning of the fetus necessary; transfer to neonatology (group 2 and 3). b) Mother: Maternal age; parity; gestational age at glucocorticoid treatment; treatment of preterm labour; medications during pregnancy; surgery and perinatal variables; history in terms of smoking, alcohol, nicotine, marihuana, other illicit drugs; Indication for ECS (group 2 and 3).
* Psychosocial data: The following variables shall be assessed from mothers by standardized and validated questionnaires: country of birth (parents, grandparents); Socio-economic status, maternal and parental education; current job situation (no, part-time, full-time); maternal and paternal trauma history (Childhood Trauma Questionnaire - Short Form from Bernstein & Fink, 1998; Karos et al. 2014); significant life events during the pregnancy (Life Event Scale from Landolt & Vollrath, 1998); maternal and paternal subjective stress during pregnancy (Perceived Stress Scale PSS-10 from Cohen, Kamarck, & Mermelstein (1983) and Klein et al. (2016); maternal and paternal mental health both retrospectively during pregnancy and currently at the assessment points after birth: anxiety and depression by means of two modules of the Patient Health Questionnaire PHQ from Spitzer, Kroenke, & Williams (1999); posttraumatic stress disorder by means of the International Trauma Questionnaire ITQ (Cloitre et al., 2018) and the infant's temperament by means of the Infant Behaviour Questionnaire IBQ - Very Short Form by Rothbart (1981). All measures are standardized and available in validated German versions.

Statistical Analyses: Aim 1 will be examined with ANCOVAs to compare total methylation / gene-expression (mRNA level) for the studied gene regions across the 3 groups. The correlation between methylation levels and gene-expression will be investigated, expecting that hypermethylation induces reduced gene-expression and vice versa.

Aim 2 will be examined by (partial) correlational analyses between predictor variables and total methylation. If requirements are met, multivariate analyses will be performed.

Aim 3 will be examined with ANCOVAs comparing IBQ-scores across the three groups.

Data will not be transformed before analysis. If the data doesn't meet the requirements for the selected statistical tests, then modified tests (e.g. one-way testing) or appropriate tests (e.g. non-parametric methods) will be used.

Statistical analysis will be performed either with the program Statistical Package for Social Sciences (SPSS, Version 25) or the statistical program R. Statistical significance will be set to a significance level of α= <.05.

Sample size: According to a power-analysis calculation with the program G*Power 3.1 (Faul, Erdfelder, Buchner & Lang, 2009), the required sample size for an ANCOVA with 3 groups, an effect size of d=0.4 (small effect) and a power of .90 is n=84.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Newborns after successful fetal surgery for MMC, delivered by ECS (elective c-section) at weeks 350 - 370.

Group 2: Healthy newborns after exposure to synthetic glucocorticoids for lung maturity during pregnancy, delivered by ECS between 350 - 400 weeks, matched for child sex with group 1. This group is needed to control for the effects of sGC exposure.

Group 3: Healthy newborns, uncomplicated pregnancy, delivered at term by ECS between 360 - 390 weeks (healthy controls). Matched for child sex with group 1.

Exclusion Criteria for all 3 groups:

* Multiple pregnancies
* Apgar 5 min <=7, or significant postpartal health problems such as respiratory distress syndrome
* ph<7.15
* General anaesthesia for ECS
* Insufficient knowledge of German or English by the mother
* Mother exposed to traumatic stress during pregnancy (other than fetal surgery)
* Non-Caucasian origin
* Egg donation

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include newborns after fetal surgery for MMC at the University Hospital Zurich and two control groups. One including healthy newborns and another including newborns after prenatal exposure to synthetic glucocorticoids (sGC) in pregnancy. Each group shall include n=30 newborns (i.e. total number of study participants: n=90). In the following paragraph you can find a detailed description of the groups as well as the inclusion and exclusion criteria for all groups.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Methylation status at NRC3C1 and the FKBP5 gene | Day 2 - Day 3
  Saliva DNA will be isolated using prepIT.L2P following manufacturer's protocol (PT-L2P; DNA Genotek Inc.). DNA concentration, A260/A280 and A260/A230 ratios for integrity and quality will be measured using the NanoDrop spectrophotometer (ThermoFisher, Switzerland).
  DNA methylation specific analysis for each selected gene (NR3C1 and FKBP5) will be conducted using the EpiTect Methyl II PCR assays (Qiagen) following the manufacturer's protocol.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ) | Week 6 and month 3
  Maternal and paternal mental health will be assessed by the Patient Health Questionnaire (PHQ) bei Spitzer et al., 1999. The questionnaire consists of 9 items with a Likert Scale from 0-3. The sum score (range 0-27) will be used. Higher scores represent more mental health problems.

OTHER OUTCOMES:
Infant Behavior Questionnaire (IBQ-Very Short Form) | Month 3
  Child temperament will be assessed by the mother-rated Infant Behavior Questionnaire (Rothbart, 2000). We will use the Very Short Form (IBQ-Very Short Form) that consists of 36 items with a Likert scale from 1-7. The 36 items can be assigned to three scales: surgency, negative affect, and effortful control. Scale scores will be computed according to the manual.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Landolt, PhD, Principal Investigator — University Children's Hospital, Zurich; Edna Gruenblatt, PhD, Principal Investigator — University of Zurich, Department of Child and Adolescent Psychiatry; Ueli Moehrlen, MD, Principal Investigator — University Children's Hospital, Zurich; Tilo Burckhart, MD, Principal Investigator — University of Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided